CLINICAL TRIAL: NCT06354075
Title: Evaluation of Patient Information in Interventional Radiology
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN302024/CHUSTE
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Patient Satisfaction
Keywords: Patient information; pediatrics; consultation; information sheet; questionnaire; interventional radiology; video; cementoplasty
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient who receives a consultation before an interventional procedure: Any patient who receives a consultation before an interventional procedure will be included. Questionary will be administrated.
  Interventions: Other: Questionary

INTERVENTIONS:
Other: Questionary — Questionary will be administrated to evaluated the information for patients on interventional radiology (explanatory video, information form, etc.).

SUMMARY:
Interventional radiology is developing. Patient information modalities are also evolving, in particular information videos.

DETAILED DESCRIPTION:
The aim of our work is therefore the evaluation of patient information in interventional radiology.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving a consultation prior to a cementoplasty procedure and children receiving a consultation prior to any interventional radiology procedure.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving a consultation prior to a cementoplasty procedure and children receiving a consultation prior to any interventional radiology procedure.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
to evaluate satisfaction of patient of explanatory videos in interventional radiology | Year : 2
  Analysis results of questionary.
To evaluate satisfaction of patient of comic book in interventional radiology | Year : 2
  Analysis results of questionary.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain GRANGE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No